CLINICAL TRIAL: NCT04854395
Title: The Effect of the Popliteal Plexus Block on Postoperative Opioid Consumption, Pain, Muscle Strength and Mobilization After Total Knee Arthroplasty - a Randomized, Controlled, Blinded Study
Brief Title: Femoral Triangle Block With Popliteal Plexus Block Versus Femoral Triangle Block Versus Adductor Canal Block for TKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regionshospitalet Silkeborg (Other)
Responsible Party: Principal Investigator, Johan Kløvgaard Sørensen, Specialist Registrar, Regionshospitalet Silkeborg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Protocol_PPB_TKA_16032021; 2021-000242-17 (EudraCT Number)
Record Dates: First submitted 2021-04-18; First posted 2021-04-22 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Pain, Acute; Opioid Use; Analgesia
MeSH Terms: conditions — Acute Pain; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Patients assigned for total knee arthroplasty are randomized into one of the three study groups in accordance to a computer-generated block randomization list in a 1:1:1 ratio (each block containing 15 numbers). Prior to surgery the patients receive the peripheral nerve blocks allocated to the group/arm they belong to:
  Group A: FTB (active) + ACB (sham) + PPB (active) Group B: FTB (active) + ACB (sham) + PPB (sham) Group C: FTB (sham) + ACB (active) + PPB (sham)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Three unblinded anesthesiologists, including the sponsor, are responsible for performing the peripheral nerve block and will not be involved in any clinical assessments, data collection or interpretation of adverse events.
  During the nerve block procedure, an opaque cloth hung over the stomach level, prevents the patient for monitoring block procedure and the ultrasound monitor. All patients experience three needle insertions in the skin (one for PPB, one for FTB incl. IFCN and one for ACB). The same time is used for each needle insertion, regardless of injection of active drug (active nerve block) or simulation of injection (sham block). Most patient are sensible to the needle insertion but are not able to feel the injection of local anesthetics. All this will ensure that the patient is blinded.
  None of the blinded outcome assessors, including primary investigator, are present during the opening of the randomization or during the nerve block procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A: Active FTB + Active PPB + Sham ACB (Active Comparator): Single shot bolus of 10 ml Marcain 5 mg/ml is used for FTB, 5 ml Marcain 5 mg/ml for IFCN + 10 ml Marcain 5 mg/ml is used for PPB
  Interventions: Drug: Marcain 5 mg/ml
- Group B: Active FTB + Sham PPB + Sham ACB (Active Comparator): Single shot bolus of 10 ml Marcain 5 mg/ml is used for FTB, 5 ml Marcain 5 mg/ml is used for IFCN
  Interventions: Drug: Marcain 5 mg/ml
- Group C: Sham FTB + Sham PPB + Active ACB (Active Comparator): Single shot bolus of 25 ml Marcain 5 mg/ml is used for ACB
  Interventions: Drug: Marcain 5 mg/ml

INTERVENTIONS:
Drug: Marcain 5 mg/ml — Total volumes of Marcain differs in each arm, depending on which nerve blocks the patients is randomized to receive. Sham block does not include injection of placebo saline, due to the risk of hydrodissection between the anatomical sections which may erase the isolation of the different nerve blocks. Instead the sham block include imitation of the real nerve block, including correct placement of the needle on the target for the block.

SUMMARY:
In this study we wish to investigate the analgesic effect 3 different nerve block regimes in patients following primary total knee arthroplasty (TKA). All nerve blocks were performed as single shot blocks with the administration of Marcain 5 mg/ml.

Regime A: proximal Femoral Triangle Block (FTB) with 10 ml including Intermediate Femoral Cutaneous Nerve Block (IFCNB) with 5 ml + Popliteal Plexus Block (PPB) with 10 ml.

Regime B: proximal FTB with 10 ml including IFCNB with 5 ml.

Regime C: Adductor Canal Block (ACB) with 25 ml.

DETAILED DESCRIPTION:
The Adductor Canal Block (ACB) is frequently used after TKA, but it is limited to provide anesthesia from the anteromedial part of the knee region. The proximal Femoral Triangle Block (FTB) is also used for TKA, and also limited to provide anesthesia from the anterior medial part of the knee joint. The FTB anesthetize the saphenus nerve, the nerve to vastus medialis, and may anesthetize the medial femoral cutaneous nerve which innervates the distal medial thigh as well as the anteromedial knee region. We included the Intermediate Femoral Cutaneous Nerve block (IFCNB) in the FTB, as the nerves can be targeted in the subcutis on the anterior thigh and easily be anesthetized during the same procedure as FTB. IFCNB anesthetize the distal anterior thigh, which may include the proximal part of the surgical incision for TKA. In the following text the proximal FTB including IFCNB will be refered as "FTB" and the dose of 15 ml will refer to 10 ml for the proximal FTB and 5 ml used for the IFCNB.

A new nerve block technique, called Popliteal Plexus Block (PPB), is specifically designed to anaesthetize nerves involved in innervation of the back of the knee joint. The analgesic effect of PPB has not yet been evaluated in randomized, controlled, blinded trials. In order to optimize pain treatment for primary TKA by improving the pain-relieving effect of peripheral nerve blocks, we aim to evaluate the analgesic effects of three different nerve block regimens (FTB + PPB versus FTB versus ACB) after primary unilateral TKA. Our outcomes include postoperative pain scores, opioid consumption, muscle strength and mobilization.

Our hypothesis is that the combination of FTB + PPB provides superior postoperative pain treatment after TKA in comparison to both FTB or ACB. The combination of FTB + PPB will reduce opioid consumption (primary outcome) and postoperative pain scores without reducing muscle strength or impairing mobilization.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo primary total knee arthroplasty in spinal anesthesia
* Able to perform a Timed Up and Go (TUG) test
* Age > 50 years old
* Ability to give their written informed consent to participating in the study after having fully understood the contents of the study
* American Society of Anesthesiologists (ASA) physical status 1, 2, or 3

Exclusion Criteria:

* Patients who cannot cooperate
* Patients who cannot understand or speak Danish.
* Patients with allergy or intolerance to the medicines used in the study
* Patients with a daily intake of strong opioids (morphine, oxycodone, ketobemidone, methadone, fentanyl)
* Patients suffering from alcohol and/or drug abuse - based on the investigator's assessment
* BMI > 40
* Diagnosed with chronic central or peripheral neurodegenerative disorders

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption in each group, A, B and C | from time of skin closure (end of surgery) until 24 hours postoperative
  Total opioid consumption is the aggregate of the opioid administered by the Patient Controlled Analgesia (PCA) pump and any potential rescue opioids administered, calculated as IV morphine equivalents

SECONDARY OUTCOMES:
Total opioid consumption in each group, A, B and C | from time of skin closure (end of surgery) until 12 hours postoperative
  Total opioid consumption is the aggregate of the opioid administered by the PCA pump and any potential rescue opioids administered, calculated as IV morphine equivalents
Post-block Maximum Voluntary Isometric Contraction (MVIC) by knee extension, calculated as a percentage of the Pre-block baseline value | A 60 minutes interval is between pre-block and post-block MVIC assessments
  Both MVIC test are assessed preoperative, using a handheld dynamometer
Post-block MVIC by ankle plantarflexion, calculated as a percentage of the Pre-block baseline value | A 60 minutes interval is between pre-block and post-block MVIC assessments
  Both MVIC test are assessed preoperative, using a handheld dynamometer
Post-block MVIC by ankle dorsiflexion, calculated as a percentage of the Pre-block baseline value | A 60 minutes interval is between pre-block and post-block MVIC assessments
  Both MVIC test are assessed preoperative, using a handheld dynamometer
Muscle strength of knee extension, graded by Manual Muscle Test (MMT) | Assessed pre-block, post-block (60 minutes after pre-block) and postoperative 5 hours after time of skin closure (end of surgery)
  Grade 3: Able to extend the knee in active Range of Motion (ROM) against gravity, Grade 2: Patient is lying on the side, with knee resting on the bed, able to extend the knee in active ROM with minimal assistance from the investigator, Grade 1: Muscle contraction of the quadriceps muscle is palpable or observable but the knee does not extend, Grade 0: No muscle contraction of the quadriceps muscle is palpable or observable
Muscle strength of ankle plantarflexion, graded by MMT | Assessed pre-block, post-block (60 minutes after pre-block) and postoperative 5 hours after time of skin closure (end of surgery)
  Grade 3: Able to plantarflex in active ROM, Grade 2: Patient is lying on the side, with ankle resting on the bed, able to plantarflex the ankle in active ROM with minimal assistance from the investigator, Grade 1: Muscle contraction of the gastrocnemius muscle is palpable or observable but the ankle does not plantarflex, Grade 0: No muscle contraction of the gastrocnemius muscle is palpable or observable
Muscle strength of ankle dorsiflexion, graded by MMT | Assessed pre-block, post-block (60 minutes after pre-block) and postoperative 5 hours after time of skin closure (end of surgery)
  Grade 3: Able to dorsiflex in active ROM Grade 2: Patient is lying on the side, with ankle resting on the bed, able to dorsiflex the ankle in active ROM with minimal assistance from the investigator, Grade 1: Muscle contraction of the tibialis anterior muscle is palpable or observable but the ankle does not dorsiflex, Grade 0: No muscle contraction of the tibialis anterior muscle is palpable or observable
Timed Up and Go (TUG) test postoperative | Assessed 5 hours after time of skin closure (end of surgery)
  Measure of seconds it takes a patient to get up from a chair with armrest, walk a distance of three meters, turn around, walk back and sit down again. All patients must use crutches for the test. If patient cannot mobilize with crutches, the test will not be performed.
Worst pain during TUG | Assessed at the end og the TUG test, 5 hours after time of skin closure (end of surgery)
  Patient will be asked to indicate worst pain, Numeric Rating Scale (NRS), 0-10, experienced during the TUG test
Pain at rest | preoperative (preblock baseline), 2, 5 (prior to TUG test), 7, 20 and 24 hours after time of skin closure (end of surgery)
  Patient will be asked to indicate pain intensity at rest (NRS, 0-10)
Pain during 90 degrees active flexion of the knee | preoperative (preblock baseline), 2, 5 (prior to TUG test), 7, 20 and 24 hours after time of skin closure (end of surgery)
  Patient will be asked to indicate worst pain intensity during active flexion of the knee towards 90 degrees (NRS, 0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Runge, PhD, Principal Investigator — Region Hospital Silkeborg
Locations (1):
- Johan Kløvgaard Sørensen, Skanderborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after acceptance from the The Danish Data Protection Agency
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At the end of study analysis
Access Criteria: Permission by investigators